CLINICAL TRIAL: NCT07249528
Title: Voice as a Digital Biomarker of Neurotoxicity in CAR T-Cell Therapy
Brief Title: A Study of Voice as a Way to Monitor for Side Effects in People Receiving CAR T-Cell Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-317
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non-hodgkin Lymphoma; Multiple Myeloma
Keywords: Non-hodgkin Lymphoma; Multiple Myeloma; Memorial Sloan Kettering Cancer Center; 25-317
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants diagnosed with non-Hodgkin lymphoma or multiple myeloma (Experimental): Participants must have pathologically confirmed Diagnosed with non-Hodgkin lymphoma or multiple myeloma.
  Interventions: Diagnostic Test: Audio Tasks

INTERVENTIONS:
Diagnostic Test: Audio Tasks — Voice recordings will be collected at baseline (pre-infusion), twice daily from Day 0 through Day +10, and, if ICANS develops, twice daily until three days after clinical resolution. A final voice recording will also be performed on Day +30

SUMMARY:
The purpose of this study is to collect voice recordings and nervous system (neurologic) assessments from people with non-Hodgkin lymphoma (NHL) or multiple myeloma (MM) who are receiving standard treatment with CAR T-cell therapy. Researchers will study whether these voice recordings and assessments are a practical (feasible) way to monitor for immune effector cell-associated neurotoxicity syndrome (ICANS). Feasibility will be measured by tracking how many participants join the study and complete the assessments.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of Disease

  o Patients must have pathologically confirmed Diagnosed with non-Hodgkin lymphoma or multiple myeloma.
* Definition of treatment and ability

  * Scheduled to receive an FDA-approved CAR-T product: Axi-cel, Liso-cel, Tisa-cel, Ide-cel, Cilta-cel, or Brexu-cel.
  * Ability to comply with twice daily voice recordings or daily neurologic assessments, as determined by the investigator.
* Age ≥ 18
* ECOG Performance Status of ≤ 2
* Required

  * Perform twice daily voice recordings using a smartphone.
  * Undergo daily neurologic assessments (e.g., ICE score, tremor evaluation).
  * Smartphone ownership.
  * Sufficient English proficiency to complete structured voice tasks in the study application.
* Comorbid Conditions

  * No pre-existing neurological conditions that significantly impair speech, including but not limited to severe dysarthria, expressive aphasia, or neurodegenerative disorders.
  * No history of significant speech or voice disorders, including laryngeal paralysis, severe dysphonia, or recent vocal cord surgery or radiation to the area.
  * No pathology affecting the vocal cords that could interfere with voice analysis, such as vocal cord paralysis, chronic laryngitis, vocal cord nodules, polyps, granulomas, or malignancies.
  * No severe hearing impairment that would interfere with voice assessments
* Language o Proficiency in spoken English is required, without the need for native-level fluency. This ensures participants can accurately perform structured voice tasks, as the application and underlying acoustic models are currently validated only in English, despite the limitation in generalizability. Participants with language barriers that prevent reliabletask completion or data interpretation will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of daily voice recordings collected | 30 days after baseline
  To prospectively collect and curate a dataset of twice daily smartphone-based voice recordings and daily neurocognitive assessments from patients undergoing CAR T-cell therapy.
Number of neurocognitive assessments collected | 30 days after baseline
  To prospectively collect and curate a dataset of twice daily smartphone-based voice recordings and daily neurocognitive assessments from patients undergoing CAR T-cell therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Roni Shouval, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering at Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Weill Cornell Medical Center (Data Analysis Only), New York, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org